CLINICAL TRIAL: NCT00619515
Title: Prospective Evaluation of Cyberknife Stereotactic Radiosurgery for Low and Low/Intermediate Risk Prostate Cancer
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Prematurely terminated at institution request
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE13807; P30CA043703 (NIH); CASE13807 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-02-20; First posted 2008-02-21 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyberKnife® stereotactic radiosurgery (Experimental)
  Interventions: Other: questionnaire administration; Procedure: implanted fiducial-based imaging; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Other: questionnaire administration — Patients complete 4 questionnaires at baseline and periodically during study to assess acute and late toxicities and quality of life (e.g., overall health status, patient function, sexual function, and urinary symptoms).
Procedure: implanted fiducial-based imaging — Undergo fiducial placement imaging
Radiation: stereotactic radiosurgery — Patients undergo fiducial placement using ultrasound. At least 5-10 days later, patients undergo CyberKnife® stereotactic radiosurgery once daily for 5 days.

SUMMARY:
RATIONALE: Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This trial is studying the side effects of stereotactic radiation therapy and to see how well it works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate in both low- and low-to-intermediate-risk groups of patients with prostate cancer, the rate of acute toxicities observed during the 5 years following CyberKnife® stereotactic radiosurgery (SRS).

Secondary

* To estimate the rate of late grade 3-5 toxicities after SRS in these patients.
* To measure biochemical disease-free survival of patients treated with this therapy.
* To measure rates of local failure, distant failure, disease-free survival, disease-specific survival, and overall survival of patients treated with this therapy.
* To measure quality of life in generic and organ-specific domains in patients treated with this therapy.
* To evaluate imaging modalities and their potential role in the detection of prostate cancer persistence, recurrence, and/or progression in patients treated with this therapy.

OUTLINE: Patients are stratified according to risk group (low risk vs low/intermediate risk).

Patients undergo fiducial placement using ultrasound. At least 5-10 days later, patients undergo CyberKnife® stereotactic radiosurgery once daily for 5 days.

Patients complete 4 questionnaires at baseline and periodically during study to assess acute and late toxicities and quality of life (e.g., overall health status, patient function, sexual function, and urinary symptoms).

After completion of study therapy, patients are followed for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Disease confirmed by biopsy within 1 year of study entry
  * Gleason score 2-7(3+4)
  * Clinical stage T1a or T2b, N0 or NX, M0 or MX

    * T- stage and N-stage determined by physical exam and available imaging studies (i.e., ultrasound, CT scan, and/or MRI)
    * M-stage determined by physical exam, CT scan, and/or MRI

      * Bone scan is not required unless clinical findings suggest possible osseous metastases
* PSA ≤ 10 ng/mL within the past 60 days
* At risk for recurrence, as defined by 1 of the following risk groups:

  * Low-risk, defined by the following combination:

    * Stage T1a-T2a, Gleason 2-6, and PSA ≤ 10 ng/mL
  * Low- to-Intermediate-risk, defined by either of the following combinations:

    * Stage T2b, Gleason 2-6, and PSA ≤ 10 ng/mL
    * Stage T2b, Gleason 3+4=7, and PSA ≤ 10 ng/mL
* Prostate volume must be ≤ 100 cc

  * Determined by measurement from CT scan or ultrasound within the past 90 days or within the past 14 days if hormone therapy is given

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion

PRIOR CONCURRENT THERAPY:

* No prior definitive therapy for prostate cancer, including prostatectomy, cryotherapy, or radiotherapy to the prostate or lower pelvis
* No more than 6 months of hormone ablation for gland downsizing

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-12; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee E. Ponsky, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - UH-Westlake, Westlake, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Started | 73
Completed | 0
Not Completed | 73
Not completed — Study Termination by IRB | 73

BASELINE CHARACTERISTICS:
Population: The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3-5 Adverse Events as Assessed by NCI CTCAE v3.0
Description: This study's primary goal is to determine the rate of acute grade 3-5 toxicities following CyberKnife treatment. Per RTOG/ECOG, acute toxicity will be defined as occurring within 90 days of completing treatment.
Time Frame: Within 90 days of completing treatment
Population: The study was terminated prematurely by the IRB due to compliance issues. As per the IRB determination, data are not accessible to the study team for reporting.
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Late Grade 3-5 Toxicities as Assessed by NCI CTCAE v3.0
Description: Late toxicity will be defined as toxicity occurring more than 90 days after treatment. It is graded based on Common Terminology Criteria for Adverse Events (CTCAE) v3.0, and RTOG/ECOG definitions.
Time Frame: Within 5 years of completing treatment
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

3. Secondary Outcome: Biochemical Disease-free Survival
Description: PSA
Time Frame: Assessed at months 3,6,12,18,24 and every 6 months through 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Disease-free Survival (Phoenix and ASTRO Definitions)
Time Frame: Assessed yearly for 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease-specific Survival
Time Frame: Assessed yearly for 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Time Frame: Assessed yearly for 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of Local Failure
Time Frame: Assessed at months 3,6,12,18,24 and every 12 months through 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

8. Secondary Outcome: Rate of Distant Failure
Time Frame: Assessed at months 3,6,12,18,24 and every 12 months through 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

9. Secondary Outcome: Quality of Life as Measured by the Short Form-12 Health Survey, Expanded Prostate Cancer Index Composite, and the American Urological Association Symptom Index, and the Utilization of Sexual Medications/Devices
Time Frame: Survey at 1,6,12 months and yearly up to 5 years
Population: as for outcome 1
Arm/Group | CyberKnife® Stereotactic Radiosurgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.
Description: The study was terminated prematurely by the IRB. As per the IRB determination, data are not accessible to the study team for reporting.
Arm/Group | CyberKnife® Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the IRB due to compliance issues. As per the IRB determination, data are not accessible to the study team for reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes